CLINICAL TRIAL: NCT03602599
Title: Natural History of Chronic Graft-versus-Host Disease in the Oral Cavity of Patients Following Allogeneic Hematopoietic Stem Cell Transplant and Including Healthy Controls
Brief Title: Chronic Graft-versus-Host Disease in the Oral Cavity of Patients Following Allogeneic Hematopoietic Stem Cell Transplant and Including Healthy Controls
Status: Recruiting | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180121; 18-D-0121
Record Dates: First submitted 2018-07-26; First posted 2018-07-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Graft Versus Host Disease
Keywords: Mouth; Alloimmunity; Autoimmunity; Salivary Gland; Ulcer; Natural History
MeSH Terms: conditions — Graft vs Host Disease; Autoimmune Diseases; Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy-controls Longitudinal Cohort: ( Cohort HL ; approximate n=20) includes subjects who will participate in up to 4 study visits across 1 year.
- Healthy-controls Short-term Cohort: ( Cohort HS ; approximate n=80) will participate in a single baseline visit.
- New Transplant Cohort: ( Cohort NT ; approximate n=300) consists of patients who are scheduled to undergo allogeneic HSCT (under another protocol at the NIH).
- Prior Transplant Cohort: ( Cohort PT ; approximate n=100) consists of patients who have already undergone allogeneic HSCT.

SUMMARY:
Background:

This study follows people who have had, or will soon have, a transplant using stem cells from another person. This is known as an allogeneic hematopoietic stem cell transplant (HSCT). Graft-versus-host disease (cGVHD) can happen after HSCT. cGVHD can cause mouth problems and more serious issues. Researchers want to study changes in the mouth that might indicate cGVHD.

Objective:

To identify cGVHD in the mouth and better understand the development, treatment, and progress of post-transplant changes in the mouth.

Eligibility:

Adults at least 18 years old who will soon undergo HSCT or have had one in the past 3 years Healthy adults at least 18 years old

Design:

All participants will have a screening visit and baseline visit. They will last 60-90 minutes. Over these two visits, participants will have:

Medical and dental history

Dental exam.

Questions about their eating habits and general health

Blood drawn through a needle in the arm

Vital signs taken

Pictures of their mouth and lips taken

Questions about their oral health, including about pain, sensitivity, or dryness

Saliva samples taken. Participants will spit into a sterile plastic tube.

Swabs taken of the mouth and some of the saliva, plaque, and fluid from the spaces between teeth and gums.

Participants may also have:

A piece of skin taken (biopsy) from the inner lining of the cheeks

A piece of skin taken (biopsy) from the lower lip

Dental X-rays

Urine pregnancy test

Most participants will have at least 7 study visits over 3 years. They will meet with a dentist and repeat baseline tests.

DETAILED DESCRIPTION:
Background:

* Chronic graft-versus-host disease (cGVHD) is a multi-organ severe alloimmune and - autoimmune disorder that occurs after allogeneic hematopoietic stem cell transplantation (HSCT). It is characterized by immune dysregulation, immunodeficiency, impaired organ function, and decreased survival.
* Manifestations of cGVHD in the oral cavity are observed in 45-85% of cGVHD patients and include 3 components: limitation of mouth opening, oral mucosal changes (lichenoid lesions, ulceration) and salivary gland changes.
* There is an urgent need for new tools to diagnose and treat oral cGVHD. To develop targeted therapies and non-invasive methods for serial screening, an improved understanding of the clinical course and underlying mechanisms of oral cGVHD are required.

Objectives:

* Advance understanding of cGVHD pathophysiology and generate hypotheses for future cGVHD studies by tracking the longitudinal development of cGVHD in the oral cavity and transplant-related changes in the oral microenvironment.
* Leverage knowledge about the impact of transplant on the oral cavity to develop better protocols for supportive dental care, to refine clinical definitions and classifications of oral cGVHD, and to test and improve criteria and tools for clinical trials.
* Include healthy volunteer cohorts both as a direct control group for HSCT patients, and to characterize measures of interest that were not previously defined in the normal oral cavity.

Eligibility:

* Patients who are scheduled to undergo allogeneic HSCT at the National Institutes of Health (NIH) or who have already undergone allogeneic HSCT at the NIH or elsewhere.
* Healthy individuals who have not undergone transplant and are willing to undergo oral exam and sample collection will be included in a control group.
* All study subjects, including patients and healthy individuals, must be able to provide written informed consent and be willing to return to the NIH Dental Clinic for scheduled evaluations.

Design:

* This is a single site, observational study with four cohorts. There are 2 transplant cohorts: the New Transplant Cohort ("Cohort NT"; approximate n=300) consists of patients who are scheduled to undergo allogeneic HSCT (under another protocol at the NIH) and the Prior Transplant Cohort ("Cohort PT"; approximate n=100) consists of patients who have already undergone allogeneic HSCT. These Cohorts will have up to 7 regularly scheduled visits across 3 years, along with a variable number of acute-episode visits. Subjects enrolled as NT or PT, who require a subsequent transplant are eligible to be either enrolled or re-enrolled into the PT cohort to be followed for the 7 visits in 3 years. Additionally, subjects will have the opportunity to participate in optional annual follow-up visits in years 4-10 post transplant.
* The other 2 Cohorts include healthy volunteers: the Healthy-controls Longitudinal (HL) Cohort ("Cohort HL"; approximate n=20) includes subjects who will participate in up to 4 study visits across 1 year, and the Healthy-controls Short-term (HS) Cohort ("Cohort HS"; approximate n=80) will participate in a single baseline visit.
* Each visit will include collection of biologic samples, patient-reported data and clinical assessments.
* Initial statistical analysis will begin with unsupervised clustering methods and simple logistic regression to identify biomarkers important in oral cGVHD. Based upon the results of these initial analyses, more complex multivariate statistical models will be developed to both classify and predict onset of oral cGVHD. Given the hypothesisgenerating nature of this study, additional prospective statistical analysis plans will be developed in consultation with a statistician as the study progresses to address specific scientific questions.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects in Cohort NT and Cohort PT must satisfy all of the following criteria in order to participate in the study:

  * Scheduled to undergo allogeneic HSCT at the NIH (Cohort NT) or have already undergone allogeneic HSCT at the NIH or another institution (Cohort PT) and are within 3 years of most recent bone marrow transplant
  * Willing to participate in protocol evaluations including saliva collection, oral swab collection, and completion of patient-reported outcome (PRO) forms
  * Willing to return to the NIH Dental Clinic for scheduled evaluations
  * Be at least 18 years of age at screening
  * Be able to understand and provide written informed consent
* Subjects in Cohort HL and Cohort HS must satisfy all of the following criteria in order to participate in the study:

  * Willing to undergo oral exam and participate in Visit 1 protocol evaluations including saliva collection, oral swab collection and oral biopsies.
  * Be at least 18 years of age at screening
  * Be able to understand and provide written informed consent
  * Potentially be age- and/or sex-matched with a transplant patient
* Subjects in Cohort HL must additionally be willing and able to return to the NIH Dental Clinic for scheduled visits across 1 year and participate in evaluations including saliva collection, oral swab collection, and completion of PRO forms

EXCLUSION CRITERIA:

* Subjects in any Cohort will be excluded if they are pregnant, as pregnancy can have a confounding effect on the oral microbiome
* Subjects in Cohort NT may not participate in the study if, in the opinion of the NIH transplant team, participation in the protocol would not be safe or in the subject s best interest
* Subjects in Cohort PT. There are no additional exclusion criteria for subjects in this cohort.
* Subjects in Cohorts HL and Cohort HS may not participate in the study if they meet either of the following criteria:

  * Have any acute oral mucosal or dental infection requiring multiple dental appointments or specialist referral for treatment; uncontrolled chronic disease; active systemic illness; are currently undergoing orthodontic treatment; history of frequent opportunistic infection; autoimmune disease; immunosuppressive medications; or prior organ, bone marrow, or peripheral blood stem cell transplant
  * Are taking medications or are on other ongoing therapies that have a known or suspected major impact on the oral microbiome
* Subjects in Cohort HL additionally may not participate if they are planning to become pregnant within the next year or refuse to have oral biopsies.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects in Cohort NT and Cohort PT will be scheduled to undergo allogeneic hematopoietic stem cell transplant at the NIH (Cohort NT) or have already undergone allogeneic HSCT at the NIH or another institution (Cohort PT) and are within 3 years of most recent bone marrow transplant. Subjects in Cohort HL and Cohort HS will be healthy volunteers and may potentially be age- and/or sex-matched with a transplant patient participant. All subjects will be at least 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2037-03-03 (Estimated); Study Completion 2037-03-03 (Estimated)

PRIMARY OUTCOMES:
Advance understanding of chronic graft versus host disease (cGVHD) pathophysiology and generate hypotheses for future cGVHD studies by tracking the longitudinal development of cGVHD in the oral cavity. | 3 years from enrollment of last participant
  Advance understanding of chronic graft versus host disease (cGVHD) pathophysiology and generate hypotheses for future cGVHD studies by tracking the longitudinal development of cGVHD in the oral cavity.

SECONDARY OUTCOMES:
Characterize post-transplant changes in oral cavity in presence and absence of cGVHD to develop better protocols for supportive dental care, Refine clinical definitions and classifications of oral cGVHD, Characterize longitudinal changes, includ... | 3 years after enrollment of last participant
  1. Characterize post-transplant changes in the oral cavity in the presence and absence of cGVHD to develop better protocols for supportive dental care.2. Refine clinical definitions and classifications of oral cGVHD.3. Characterize longitudinal changes in the oral microbiome4. Include healthy volunteer cohorts both as a direct control group for HSCT patients, and to characterize measures of interest that were not previously defined in the normal oral cavity.5. Test and improve criteria and tools for clinical trials

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline W Mays, D.D.S., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Protocol is silent on IPD sharing.

REFERENCES:
- [Background] Mays JW, Fassil H, Edwards DA, Pavletic SZ, Bassim CW. Oral chronic graft-versus-host disease: current pathogenesis, therapy, and research. Oral Dis. 2013 May;19(4):327-46. doi: 10.1111/odi.12028. Epub 2012 Oct 28. PMID 23107104
- [Background] Cooke KR, Luznik L, Sarantopoulos S, Hakim FT, Jagasia M, Fowler DH, van den Brink MRM, Hansen JA, Parkman R, Miklos DB, Martin PJ, Paczesny S, Vogelsang G, Pavletic S, Ritz J, Schultz KR, Blazar BR. The Biology of Chronic Graft-versus-Host Disease: A Task Force Report from the National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease. Biol Blood Marrow Transplant. 2017 Feb;23(2):211-234. doi: 10.1016/j.bbmt.2016.09.023. Epub 2016 Oct 3. PMID 27713092
- [Background] Jagasia MH, Greinix HT, Arora M, Williams KM, Wolff D, Cowen EW, Palmer J, Weisdorf D, Treister NS, Cheng GS, Kerr H, Stratton P, Duarte RF, McDonald GB, Inamoto Y, Vigorito A, Arai S, Datiles MB, Jacobsohn D, Heller T, Kitko CL, Mitchell SA, Martin PJ, Shulman H, Wu RS, Cutler CS, Vogelsang GB, Lee SJ, Pavletic SZ, Flowers ME. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant. 2015 Mar;21(3):389-401.e1. doi: 10.1016/j.bbmt.2014.12.001. Epub 2014 Dec 18. PMID 25529383
- [Derived] Leinbach LI, Boroumand S, Masuch LR, Nguyen JT, Ganesan SM, Mays JW. Oral Health Characteristics 2 Years following Allogeneic Cell Transplant. J Dent Res. 2025 Sep;104(10):1061-1068. doi: 10.1177/00220345251329351. Epub 2025 May 12. PMID 40353516
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-D-0121.html